CLINICAL TRIAL: NCT01704131
Title: Pharmacokinetics of Levosimendan in Children With Acute Heart Failure
Brief Title: Levosimendan Pharmacokinetics in Children
Acronym: LevoCorKids
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Principal Investigator, Peter Paul Roeleveld, Principal Investigator, Leiden University Medical Center
Other Study IDs: ICCE12.001
Record Dates: First submitted 2012-05-23; First posted 2012-10-11 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Acute Heart Failure
Keywords: Levosimendan; Children; Pharmacokinetics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- children > 6 months: children > 6 months of age
- children < 6 months: children < 6 months

SUMMARY:
Levosimendan is a drug used in patients with heart failure and has several advantages over other heart failure drugs. A lot of research has been done with Levosimendan in Adults, and the way the body handles the drug (pharmacokinetics) and responds to the drug (pharmacodynamics) are well established. But, in children this information is lacking despite the fact that Levosimendan is increasingly used in children of all ages. The investigators aim to describe which Levosimendan dose leads to which drug levels in children of different ages.

DETAILED DESCRIPTION:
Rationale: Levosimendan, a calcium-sensitizer, is a relatively new inotropic drug with the benefit over conventional inotropes that it does not increase myocardial oxygen demand or lead to arrhythmias. Levosimendan has a relatively unique pharmacokinetic profile, after a 24 hour infusion its clinical effects remain for several days. This is achieved through the continuing haemodynamic effects of its active metabolites, which have a half life of approximately 80 hours compared to 1 hour of Levosimendan itself. Levosimendan has been extensively studied in adults and is used in ischemic heart disease, acute heart failure, chronic heart failure, following cardiac surgery, and in septic shock. Due to the inotropic properties and its strong pulmonary vasodilatory effect, Levosimendan could also be very useful as perioperative therapy in children with congenital heart disease, low cardiac output, or pulmonary artery hypertension.

Although experience with levosimendan in children is still scarce in the literature, initial reports have been promising and Levosimendan is used more and more often as a (rescue) therapy in children with heart failure. However, current dosing regimens in children are based on adult pharmacokinetic evidence. One pediatric report suggests that the pharmacokinetic profile of a single loading dose of Levosimendan is probably similar in children older than 6 months compared to adults. The pharmacokinetic profile of a 24-hour infusion of Levosimendan has not yet been studied in children. It is very important to study the pharmacokinetics of this useful drug in different age groups because of the diversity of the population due to age, volume of distribution, ontogeny of the metabolizing enzymes, and the influence of disease state on pharmacokinetics and pharmacodynamics.

Objective: To describe the pharmacokinetic profile of a 24 hour infusion of levosimendan and its active metabolites in children with acute or chronic heart failure.

Study design: Observational study of Levosimendan levels in children treated with Levosimendan because of heart failure.

Study population: Children (< 16 years) admitted to the pediatric intensive care unit, with acute or chronic heart failure.

Intervention (if applicable): no intervention Main study parameters/endpoints: The primary endpoint of the study is to describe the pharmacokinetic profile by determining plasma levels of levosimendan and its metabolites during 12 days following a 24-hour infusion in children with heart failure in different age groups. Secondary endpoints are the clinically measured hemodynamic variables (heart rate, bloodpressure, lactate, troponin, pro-BNP, venous saturation) and echocardiographic variables (ejection fraction, shortening fraction, tissue Doppler) of all patients.

ELIGIBILITY:
Inclusion Criteria:

* All children admitted to the Pediatric Intensive Care Unit with Acute Heart Failure who will receive Levosimendan as part of their treatment.

Exclusion Criteria:

* no informed consent
* no sampling line

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children admitted to the Pediatric Intensive Care Unit with Acute Heart Failure who will receive Levosimendan as part of their treatment.
  Patients will receive Levosimendan whether they participate in the study (sampling levosimendan levels) or not.
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2012-11 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
the pharmacokinetic profile of levosimendan and is metabolites | 3 years
  AUC, Cmax, half-life, steady state concentration, plasma clearance, volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: Peter P Roeleveld, MD, Principal Investigator — Leiden University Medical Center; Heleen E Bunker-Wiersma, MD, phd, Study Chair — Leiden University Medical Center
Locations (1):
- PICU Leiden University Medical Center, Leiden, Netherlands